CLINICAL TRIAL: NCT06324019
Title: Developing Gynecological Examination Dress and Determining Its Effect on Perception of Privacy and Satisfaction: Randomized Controlled Trial
Brief Title: Gynaecological Examination Gown and Patient Satisfaction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ayşegül muslu (Other)
Responsible Party: Sponsor-Investigator, ayşegül muslu, lecturer, Ege University
Organization: Ege University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Ethics number E.405221
Record Dates: First submitted 2024-02-08; First posted 2024-03-21 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Gynecology; Gynecology/Obstetrics Conditions

STUDY DESIGN:
Intervention Model Description: The study was carried out as a post-test control group design from randomised controlled studies. The intervention group of the study was dressed in gynaecological examination clothes, while the control group used the drape given to the patient during the examination, which is a routine practice in the health institution where the study was conducted.
  Hypotheses of the Study
  1. Ho: There is no difference between the perception of privacy in the experimental and control group women.
     H1: There is a difference between the perception of privacy in the experimental group and control group women.
  2. Ho: There is no difference between the perception of satisfaction in the experimental group and control group women.
  H1: There is a difference between the satisfaction perception of women in the experimental group and the control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Developing Gynecological Examination Dress (Experimental): Gown will be put on the patient before gynaecological examination and their satisfaction will be evaluated
  Interventions: Other: putting on an examination gown

INTERVENTIONS:
Other: putting on an examination gown — During the gynecological examination, the patient in the experimental group will be made to wear an examination gown, while the patient in the control group will use the routine practice of the hospital. In this way, with the gynecological examination clothing to be developed, the body privacy of the patients will be protected during the examination. In addition, women will feel less anxiety during gynecological examination and important steps will be taken in maintaining women's health by ensuring regular gynecological examination.

SUMMARY:
The attitude of the health personnel before, during and after the examination and the positive examination experience of the person have a significant impact on ensuring the continuity of the subsequent examination and increasing the quality of the service provided. The use of different clothes in the patient during the examination will ensure that the patient's physical privacy is ensured from the moment of application, during diagnosis and treatment, and that the examination experience will be positively affected by preventing the use of additional covers to protect the privacy of all patients during examination and intervention. This will contribute to the maintenance of health by eliminating the intense stress and embarrassment experienced by patients during the examination and ensuring that they regularly attend health checks. In addition, meeting the privacy expectations of the patients will ensure that they are satisfied with the health service they receive, thus increasing the quality of the health service provided.

The attitude of the health personnel before, during and after the examination and the positive examination experience of the person have an important effect on ensuring the continuity of the subsequent examination and increasing the quality of the service provided. With the examination suit, it will be ensured that the patient's bodily privacy is ensured from the moment of application, during diagnosis, treatment and care, the use of the same cover to protect the privacy of all patients during examination and intervention will be prevented to prevent infection transmission and the examination experience will be positively affected. Thus, the intense stress and embarrassment experienced by patients during the examination will be eliminated and will contribute to the maintenance of health through regular visits to health checks. In addition, meeting the privacy expectations of patients will ensure that they are satisfied with the health service they receive, thus increasing the quality of the health service provided. In order to ensure patient privacy, to protect and improve women's health and to provide convenience in gynecological examination, the gynecological examination garment to be used in the examination can be designed as disposable, perineum and thigh open for the examination to be performed. In order to protect privacy, extra parts can be used to ensure that the open parts remain closed outside the examination process. Properties of the fabric used in the examination garment;

* Grama: 32,07 g/m^2
* Explosion.: 135,77 kpç
* Detachment: Ȼ: 115NȺ: 120 N
* Air permeability: 1750
* Type of material: Polypropylene

The study was carried out as a post-test control group design from randomised controlled studies. The intervention group of the study was dressed in gynaecological examination clothes, while the control group used the drape given to the patient during the examination, which is a routine practice in the health institution where the study was conducted.

ELIGIBILITY:
Inclusion Criteria:

* Women who will undergo gynaecological examination
* Women who volunteered to participate in the study
* no physical disabilities

Exclusion Criteria:

* Women who will not undergo a gynaecological examination

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — the outfit to be developed will be given to women during gynaecological examination
Enrollment: 150 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-06-22 (Actual)

PRIMARY OUTCOMES:
Gynaecological examination gown | 1 year
  In this study, women's satisfaction with the clothing developed will be evaluated with the Body Privacy in Gynecology and Obstetrics Scale. The scale is a five-point Likert-type scale with thirty-seven items consisting of "General Privacy", "Rights and Privacy", "Ethics and Privacy" and "Clinical Privacy" sub-dimensions. All of the statements in the dimensions are positive and the answers given to each item were summed by scoring between 1-5 and then the mean values were calculated for each item. It is understood that the higher the mean scores obtained from the scale, the more sensitive the participants are about privacy in the relevant area. The General Rights and Privacy Dimension of the scale consists of statements between items 1-9. Rights and privacy dimension consists of statements between items 10-14. Ethical rights and privacy dimension consists of statements between items 15-19. Clinical and privacy dimension consists of statements between items 20-37.

CONTACTS AND LOCATIONS:
Locations (1):
- EGE, Izmir, Konak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No